CLINICAL TRIAL: NCT02193087
Title: A Randomized, Double Blind, Phase 2 Study to Assess the Safety and Immunogenicity of Three Formulations of Takeda's Tetravalent Dengue Vaccine Candidate (TDV) in Healthy Adults
Brief Title: Safety and Immunogenicity of Three Formulations of Takeda's Tetravalent Dengue Vaccine Candidate (TDV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DEN-106; U1111-1154-9746 (Other: World Health Organization)
Record Dates: First submitted 2014-07-15; First posted 2014-07-17 (Estimated); Results first posted 2016-06-29 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Dengue Fever
Keywords: Drug therapy
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A: TDV Liquid + Placebo (Active Comparator): Takeda's Tetravalent Dengue Vaccine Candidate (TDV) Liquid Formulation 1, diluted 1:5 with vaccine diluent, subcutaneous injection on Day 1, and TDV Liquid Formulation placebo-matching solution, subcutaneous injection, once on Day 90 (Month 3).
  Interventions: Drug: TDV Liquid Formulation 1; Drug: Placebo
- Group B: TDV Liquid (Active Comparator): TDV Liquid Formulation 1, diluted 1:5 with vaccine diluent, subcutaneous injection on Day 1 and Day 90 (Month 3).
  Interventions: Drug: TDV Liquid Formulation 1
- Group C: TDV Liquid (Experimental): TDV Liquid Formulation 2, subcutaneous injection on Day 1 and Day 90 (Month 3).
  Interventions: Drug: TDV Liquid Formulation 2
- Group D: TDV Lyophilized (Experimental): TDV Lyophilized Formulation reconstituted with water, subcutaneous injection on Day 1 and Day 90 (Month 3).
  Interventions: Drug: TDV IDT Lyophilized

INTERVENTIONS:
Drug: TDV Liquid Formulation 1 — TDV Liquid Formulation 1 for subcutaneous injection
  Arms: Group A: TDV Liquid + Placebo; Group B: TDV Liquid
Drug: TDV Liquid Formulation 2 — TDV Liquid Formulation 2 for subcutaneous injection
  Arms: Group C: TDV Liquid
Drug: TDV IDT Lyophilized — TDV Lyophilized Formulation for subcutaneous injection
  Arms: Group D: TDV Lyophilized
Drug: Placebo — TDV liquid formulation placebo-matching solution for subcutaneous injection
  Arms: Group A: TDV Liquid + Placebo

SUMMARY:
The purpose of this study is to evaluate the equivalence of the lyophilized formulation of Takeda's Tetravalent Dengue Vaccine Candidate (TDV) compared with the liquid formulation of TDV.

DETAILED DESCRIPTION:
The vaccine being tested in this study is Takeda's Tetravalent Dengue Vaccine Candidate (TDV). This study is designed to determine whether the lyophilized formulation provides equivalent safety and immunogenicity as the original liquid formulation. An exploratory analysis has been added for the purpose of understanding whether there is a manufacturing or formulation effect on the vaccine.

The study will enroll approximately 1000 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the four study groups-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Group A: TDV Liquid Formulation 1, subcutaneous (SC) injection on Day 1 and placebo (dummy) SC at Month 3 - this is a liquid that looks like the study drug but has no active ingredient
* Group B: TDV Liquid Formulation 1, SC injection Day 1 and Month 3
* Group C: TDV Liquid Formulation 2, SC injection Day 1 and Month 3
* Group D: TDV Lyophilized formulation SC injection Day 1 and Month 3

In order to keep the treatment arms undisclosed to the participant and the doctor, participants will receive a placebo injection at any study visit where TDV is not being administered (Month 3). Participants will be asked to record any adverse events that may be related to the vaccine or the injection in a diary card for 28 days after each vaccination.

This multi-center trial will be conducted in the United States. The overall time to participate in this study is up to 10 months. Participants will make 9 visits to the clinic including a final visit 1 month after last dose of study drug for a follow-up assessment. A follow up phone call will be done 6 months after the last dose to assess serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Is aged 18 to 49 years, at the time of enrollment inclusive.
2. Individuals who are in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs) and clinical judgment of the investigator.
3. Signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any trial procedures, after the nature of the trial has been explained according to local regulatory requirements.
4. Individuals who can comply with trial procedures and are available for the duration of follow-up.

Exclusion Criteria:

1. Febrile illness (temperature ≥ 38°C or 100.4°F) or moderate or severe acute illness or infection at the time of enrollment. Trial entry should be delayed until the illness has improved.
2. History or any illness that, in the opinion of the investigator, might interfere with the results of the trial or pose additional risk to the participants due to participation in the trial, including but not limited to: a. Known hypersensitivity or allergy to any of the vaccine components; b. Individuals with history of substance or alcohol abuse within the past 6 months; c. Female participants who are pregnant or breastfeeding; d. Individuals with any serious chronic or progressive disease according to judgment of the investigator (e.g., neoplasm, insulin dependent diabetes, cardiac, renal or hepatic disease, neurologic or seizure disorder or Guillain-Barré syndrome); e. Known or suspected impairment/alteration of immune function, including: i. Chronic use of oral steroids (equivalent to 20 mg/day prednisone ≥ 12 weeks / ≥ 2 mg/kg body weight / day prednisone ≥ 2 weeks) within 60 days prior to Day 1 (use of inhaled, intranasal, or topical corticosteroids is allowed); Receipt of parenteral steroids (equivalent to 20 mg/day prednisone ≥ 12 weeks / ≥ 2 mg/kg body weight / day prednisone ≥ 2 weeks) within 60 days prior to Day 1; iii. Administration of immunoglobulins and/or any blood products within the three months preceding the first administration of the investigational vaccine or planned administration during the trial; iv. Receipt of immunostimulants within 60 days prior to Day 1; v. Immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within 6 months preceding (first) vaccination; vi. human immunodeficiency virus (HIV) infection or HIV-related disease; vii. Genetic immunodeficiency.
3. Individuals who received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this trial or who are planning to receive any vaccine within 28 days of investigational vaccine administration.
4. Individuals participating in any clinical trial with another investigational product 30 days prior to first trial visit or intent to participate in another clinical trial at any time during the conduct of this trial.
5. Individuals who are first degree relatives of individuals involved in trial conduct.
6. If female of childbearing potential, sexually active, and has not used any of the acceptable contraceptive methods for at least 2 months prior to trial entry: a. Of childbearing potential is defined as status post onset of menarche and not meeting any of the following conditions: menopausal (for at least 2 years), bilateral tubal ligation (at least 1 year previously), bilateral oophorectomy (at least 1 year previously) or hysterectomy; b. Acceptable birth control methods are defined as one or more of the following: i. Hormonal contraceptive (such as oral, injection, transdermal patch, implant, cervical ring); ii. Barrier (condom with spermicide or diaphragm with spermicide) each and every time during intercourse; iii. Intrauterine device (IUD); iv. Monogamous relationship with vasectomized partner. Partner must have been vasectomized for at least six months prior to the participants' trial entry.
7. If female of childbearing potential, sexually active and refuses to use an acceptable contraceptive method through to 6 weeks after the last dose of investigational vaccine.
8. Individuals with body mass index (BMI) greater than or equal to 35.
9. Participants who received previous vaccination (in a clinical trial or with an approved product) against flaviviruses including dengue, yellow fever (YF), West Nile (WN), Japanese Encephalitis (JE), and St. Louis encephalitis.
10. Documented or suspected disease caused by dengue, JE, WN, YF virus, and/or St. Louis encephalitis.
11. History of travel to dengue endemic areas including the Caribbean, Mexico, Central America, South America or Southeast Asia during the 6 months prior to screening or planned travel to a dengue endemic area during the study period.
12. Clinically significant abnormality in the screening laboratory tests as judged by the Investigator.
13. History of recurring headaches or migraines (more frequent than once per week) or on prescription medication for treatment of recurring headaches or migraines.
14. Blood tests positive for antibodies to HIV-1/2, Hepatitis C and Hepatitis B surface antigen.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1002 (Actual)
Dates: Start 2014-08-06 (Actual); Primary Completion 2015-05-19 (Actual); Study Completion 2015-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (7):
- United States (7):
  - Hope Research Institute, Phoenix, Arizona
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Advanced Clinical Research, Meridian, Idaho
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Tekton Research, Austin, Texas

REFERENCES:
- [Derived] Rauscher M, Youard Z, Faccin A, Patel SS, Pang H, Zent O. Pregnancy outcomes following unintentional exposure to TAK-003, a live-attenuated tetravalent dengue vaccine. Expert Rev Vaccines. 2025 Dec;24(1):221-229. doi: 10.1080/14760584.2025.2480297. Epub 2025 Mar 27. PMID 40099800
- [Derived] Turner M, Papadimitriou A, Winkle P, Segall N, Levin M, Doust M, Johnson C, Lucksinger G, Fierro C, Pickrell P, Raanan M, Tricou V, Borkowski A, Wallace D. Immunogenicity and safety of lyophilized and liquid dengue tetravalent vaccine candidate formulations in healthy adults: a randomized, phase 2 clinical trial. Hum Vaccin Immunother. 2020 Oct 2;16(10):2456-2464. doi: 10.1080/21645515.2020.1727697. Epub 2020 Mar 2. PMID 32119591

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 7 investigative sites in the United States from 22 July 2014 to 19 May 2015.
Pre-assignment Details: Healthy volunteers were enrolled in a 2:1:1:6 ratio into 1 of 4 study groups: 1 study group received 1 dose and 3 study groups received 2 doses.
Period: Overall Study
Arm/Group | Group A: TDV Liquid + Placebo | Group B: TDV Liquid | Group C: TDV Liquid | Group D: TDV Lyophilized
Started | 199 | 100 | 100 | 603
Received Vaccination | 197 | 97 | 100 | 602
Completed | 162 | 86 | 93 | 524
Not Completed | 37 | 14 | 7 | 79
Not completed — Adverse Event | 2 | 0 | 0 | 11
Not completed — Lost to Follow-up | 14 | 6 | 4 | 37
Not completed — Protocol Violation | 2 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 10 | 3 | 1 | 19
Not completed — Other Reason Not Specified | 7 | 2 | 1 | 9
Not completed — Did Not Receive Any Vaccination | 2 | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: TDV Liquid + Placebo | Group B: TDV Liquid | Group C: TDV Liquid | Group D: TDV Lyophilized | Total
Number analyzed (Participants) | 199 | 100 | 100 | 603 | 1002
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (8.66) | 30.9 (8.72) | 34.1 (9.20) | 31.9 (8.89) | 32.1 (8.88)
Age, Customized [Number; unit: participants]
  Adults (18-64 Years) | 199 | 100 | 100 | 603 | 1002
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 51 | 47 | 298 | 505
  Male | 90 | 49 | 53 | 305 | 497
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 40 | 22 | 21 | 120 | 203
  Non-Hispanic or Latino | 152 | 75 | 76 | 464 | 767
  Not Reported | 7 | 3 | 3 | 15 | 28
  Unknown | 0 | 0 | 0 | 3 | 3
  Missing | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 4 | 2 | 1 | 8 | 15
  Asian | 5 | 1 | 3 | 16 | 25
  Black or African American | 51 | 27 | 26 | 146 | 250
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 1 | 2 | 5
  White | 125 | 66 | 69 | 408 | 668
  Multiracial | 3 | 1 | 0 | 15 | 19
  Missing | 9 | 3 | 0 | 8 | 20
Region of Enrollment [Number; unit: participants]
  United States | 199 | 100 | 100 | 603 | 1002
Height [Mean (Standard Deviation); unit: cm] | 169.55 (9.284) | 171.13 (10.466) | 169.84 (9.727) | 170.69 (9.680) | 170.42 (9.689)
Weight [Mean (Standard Deviation); unit: kg] | 76.95 (14.362) | 78.96 (16.878) | 75.96 (16.099) | 77.49 (15.649) | 77.37 (15.569)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.71 (4.180) | 26.81 (4.496) | 26.30 (5.006) | 26.53 (4.513) | 26.57 (4.494)

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer (GMT) of Neutralizing Antibodies for Each of the Four Dengue Serotypes Comparing Group D To Groups A and B Combined
Description: Geometric mean titer (GMT) of neutralizing antibodies for each of the four dengue serotypes as measured by Plaque Reduction Neutralization Test resulting in 50% reduction in Plaques (PRNT50). The four dengue serotypes are DEN-1, DEN-2, DEN-3 and DEN-4.
  A 90% Confidence Interval (CI) for the ratio of GMT (or equivalently the difference of the log transformed GMT) was provided, for each serotype, for the comparison of the lyophilized formulation (Group D) versus the liquid formulation 1 (Groups A+B combined). An Analysis of Variance (ANOVA) model for the natural log-transformed GMT at month 1 with study group as a factor was used for analysis.
Time Frame: Month 1
Population: Per-Protocol Set (PPS) included all randomized participants who received the planned number of investigational vaccine doses, had serology data at Baseline and Month 1 and had no major protocol violations. Participants seropositive at Baseline are not included.
Measure: Least Squares Mean (90% Confidence Interval); unit: titer
Groups:
- Group A + Group B Combined: Group A: Takeda's Tetravalent Dengue Vaccine Candidate (TDV) Liquid Formulation 1, diluted 1:5 with vaccine diluent, subcutaneous injection on Day 1, and TDV Liquid Formulation placebo-matching solution, subcutaneous injection, once on Day 90 (Month 3).
  Group B: TDV Liquid Formulation 1, diluted 1:5 with vaccine diluent, subcutaneous injection on Day 1 and Day 90 (Month 3).
Arm/Group | Group A + Group B Combined | Group D: TDV Lyophilized
Number analyzed (Participants) | 220 | 454
titer
  DEN-1 | 635.04 [530.62 to 760.00] | 181.23 [159.92 to 205.37]
  DEN-2 | 15104.68 [13135.48 to 17369.09] | 16072.59 [14583.29 to 17713.99]
  DEN-3 | 186.32 [151.11 to 229.74] | 272.75 [235.75 to 315.57]
  DEN-4 | 88.87 [72.29 to 109.25] | 65.67 [56.88 to 75.82]
Statistical Analysis 1: Comparison: Group A + Group B Combined vs Group D: TDV Lyophilized; DEN-1; Test type: Non-Inferiority or Equivalence — Based on the Two One-Sided Tests (TOST) with α=0.05, if the 90% CI for the ratio of GMT for a given dengue serotype for the comparison was within the range of 0.67 and 1, then the 2 formulations were deemed equivalent; LS Mean Ratio = 0.29, 90% CI 2-sided [0.23 to 0.36]
Statistical Analysis 2: Comparison: Group A + Group B Combined vs Group D: TDV Lyophilized; DEN-2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; LS Mean Ratio = 1.06, 90% CI 2-sided [0.90 to 1.26]
Statistical Analysis 3: Comparison: Group A + Group B Combined vs Group D: TDV Lyophilized; DEN-3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; LS Mean Ratio = 1.46, 90% CI 2-sided [1.13 to 1.89]
Statistical Analysis 4: Comparison: Group A + Group B Combined vs Group D: TDV Lyophilized; DEN-4; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; LS Mean Ratio = 0.74, 90% CI 2-sided [0.57 to 0.95]

2. Secondary Outcome: Geometric Mean Titers (GMT) of Neutralizing Antibodies for Each of the Four Dengue Serotypes Comparing Group D With Group B
Description: Geometric mean titer (GMT) of neutralizing antibodies for each of the four dengue serotypes as measured by Plaque Reduction Neutralization Test resulting in 50% reduction in Plaques (PRNT50). The four dengue serotypes are DEN-1, DEN-2, DEN-3 and DEN-4. ANOVA model for the natural log-transformed GMT at month 1 with study group as a factor was used for analysis.
Time Frame: Months 1 and 4
Population: PPS included all randomized participants who received the planned number of investigational vaccine doses, had serology data at Baseline and Month 1 and had no major protocol violations. Participants seropositive at Baseline are not included. "n" in each of the categories is the number of participants with data available at the given time-point.
Measure: Least Squares Mean (90% Confidence Interval); unit: titer
Arm/Group | Group B: TDV Liquid | Group D: TDV Lyophilized
Number analyzed (Participants) | 74 | 454
titer
  Month 1 DEN-1 (n=74, 454) | 627.56 [458.91 to 858.18] | 181.23 [159.71 to 205.63]
  Month 1 DEN-2 (n=74, 454) | 17876.66 [14186.79 to 22526.23] | 16072.59 [14640.33 to 17644.97]
  Month 1 DEN-3 (n=74, 454) | 220.29 [154.23 to 314.64] | 272.75 [236.19 to 314.98]
  Month 1 DEN-4 (n=74, 454) | 88.25 [62.10 to 125.43] | 65.67 [56.98 to 75.68]
  Month 4 DEN-1 (n=73, 435) | 267.80 [205.46 to 349.06] | 113.43 [101.76 to 126.44]
  Month 4 DEN-2 (n=73, 435) | 4160.29 [3508.92 to 4932.58] | 3772.95 [3518.74 to 4045.53]
  Month 4 DEN-3 (n=73, 435) | 106.98 [85.08 to 134.52] | 132.73 [120.84 to 145.79]
  Month 4 DEN-4 (n=73, 435) | 31.56 [24.82 to 40.14] | 28.84 [26.13 to 31.82]

3. Secondary Outcome: Percentage of Participants With a Seropositive Response for Each of the Four Dengue Serotypes Comparing Group D With Groups A and B Combined
Description: A seropositive response is defined as a reciprocal neutralizing titer ≥ 10. The four dengue serotypes are DEN-1, DEN-2, DEN-3 and DEN-4.
Time Frame: Month 1
Population: Per-Protocol Set (PPS) included all randomized participants who received the planned number of investigational vaccine doses, had serology data at Baseline and Month 1, and have no major protocol violations. Participants seropositive at Baseline are not included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Group A + Group B Combined: Group A: TDV Liquid Formulation 1, diluted 1:5 with vaccine diluent, subcutaneous injection on Day 1, and TDV Liquid Formulation placebo-matching solution, subcutaneous injection, once on Day 90 (Month 3).
  Group B: TDV Liquid Formulation 1, diluted 1:5 with vaccine diluent, subcutaneous injection on Day 1 and Day 90 (Month 3).
Arm/Group | Group A + Group B Combined | Group D: TDV Lyophilized
Number analyzed (Participants) | 220 | 454
percentage of participants
  DEN-1 | 97.7 [94.8 to 99.3] | 93.6 [91.0 to 95.7]
  DEN-2 | 100.0 [98.3 to 100.0] | 99.6 [98.4 to 99.9]
  DEN-3 | 91.8 [87.4 to 95.1] | 93.4 [90.7 to 95.5]
  DEN-4 | 80.9 [75.1 to 85.9] | 80.0 [76.0 to 83.5]

4. Secondary Outcome: Percentage of Participants With a Seropositive Response for Each of the Four Dengue Serotypes Comparing Group D With Group B
Description: as for outcome 3
Time Frame: Months 1 and 4
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group B: TDV Liquid | Group D: TDV Lyophilized
Number analyzed (Participants) | 74 | 454
percentage of participants
  Month 1 DEN-1 (n=74, 454) | 97.3 [90.6 to 99.7] | 93.6 [91.0 to 95.7]
  Month 1 DEN-2 (n=74, 454) | 100.0 [95.1 to 100.0] | 99.6 [98.4 to 99.9]
  Month 1 DEN-3 (n=74, 454) | 95.9 [88.6 to 99.2] | 93.4 [90.7 to 95.5]
  Month 1 DEN-4 (n=74, 454) | 78.4 [67.3 to 87.1] | 80.0 [76.0 to 83.5]
  Month 4 DEN-1 (n=73, 435) | 97.3 [90.5 to 99.7] | 98.2 [96.4 to 99.2]
  Month 4 DEN-2 (n=73, 435) | 100.0 [95.0 to 100.0] | 100.0 [99.1 to 100.0]
  Month 4 DEN-3 (n=73, 435) | 98.6 [92.6 to 100.0] | 98.9 [97.3 to 99.6]
  Month 4 DEN-4 (n=73, 435) | 83.6 [73.0 to 91.2] | 79.3 [75.2 to 83.0]

5. Secondary Outcome: Percentage of Participants With Solicited Local (Injection Site) Adverse Events (AEs)
Description: Solicited local AEs at injection site are defined as pain, erythema and swelling that occurred at least once within 7 days after either vaccination, as recorded by the participants in a diary. Percentages are based on the number of participants with diary data available.
Time Frame: Days 1 through 7 after each vaccination
Population: Participants from the Safety Set (SS) with evaluable data and who received at least 1 dose of study vaccine (or placebo), including a partial dose. "n" in each of the categories is the number of participants with data available for analysis.
Measure: Number; unit: percentage of participants
Groups:
- Group A and Group B Combined: Group A: Takeda's Tetravalent Dengue Vaccine Candidate (TDV) Liquid Formulation 1, diluted 1:5 with vaccine diluent, subcutaneous injection on Day 1, and TDV Liquid Formulation placebo-matching solution, subcutaneous injection, once on Day 90 (Month 3).
  Group B: TDV Liquid Formulation 1, diluted 1:5 with vaccine diluent, subcutaneous injection on Day 1 and Day 90 (Month 3).
Arm/Group | Group A: TDV Liquid + Placebo | Group B: TDV Liquid | Group A and Group B Combined | Group C: TDV Liquid | Group D: TDV Lyophilized
Number analyzed (Participants) | 191 | 95 | 294 | 99 | 583
percentage of participants
  Pain (n=191, 95, 99, 583) | 43.5 | 48.4 | 45.1 | 51.5 | 45.3
  Erythema (n=191, 95, 99, 582) | 35.6 | 41.1 | 37.4 | 51.5 | 43.0
  Swelling (n=191, 95, 99, 582) | 11.5 | 20.0 | 14.3 | 24.2 | 21.6

6. Secondary Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs)
Description: Solicited systemic AEs are defined as asthenia, fever, headache, malaise, and myalgia that occurred at least once within 14 days after either vaccination, as recorded by the participants in a diary. Percentages are based on the number of participants with diary data available.
Time Frame: Days 1 through 14 after each vaccination
Population: Participants from the SS with evaluable data and who received at least 1 dose of study vaccine (or placebo), including a partial dose.
Measure: Number; unit: percentage of participants
Arm/Group | Group A: TDV Liquid + Placebo | Group B: TDV Liquid | Group C: TDV Liquid | Group D: TDV Lyophilized
Number analyzed (Participants) | 191 | 95 | 99 | 584
percentage of participants
  Headache | 40.8 | 43.2 | 38.4 | 41.1
  Asthenia | 27.7 | 23.2 | 25.3 | 26.9
  Malaise | 29.3 | 27.4 | 25.3 | 25.3
  Myalgia | 30.4 | 38.9 | 30.3 | 33.2
  Fever (≥38 °C) | 1.6 | 3.2 | 1.0 | 1.7

7. Secondary Outcome: Percentage of Participants With Solicited Local (Injection Site) Adverse Events (AEs) by Severity
Description: The percentage of participants with solicited local AEs at injection site of varying severity are reported. Solicited local AEs are defined as pain, erythema and swelling that occurred at least once within 7 days after either vaccination, as recorded by the participants in a diary. Participants with multiple episodes are categorized using the highest severity level. Percentages are based on the number of participants with diary data available.
Time Frame: Days 1 through 7 after each vaccination
Population: Participants from the SS with evaluable data and who received at least 1 dose of study vaccine (or placebo), including a partial dose. "n" in each of the categories is the number of participants with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Group A: TDV Liquid + Placebo | Group B: TDV Liquid | Group C: TDV Liquid | Group D: TDV Lyophilized
Number analyzed (Participants) | 191 | 95 | 99 | 583
percentage of participants
  Pain_Mild (n=191, 95, 99, 583) | 34.6 | 36.8 | 41.4 | 34.8
  Pain_Moderate (n=191, 95, 99, 583) | 6.8 | 8.4 | 8.1 | 9.3
  Pain_Severe (n=191, 95, 99, 583) | 2.1 | 3.2 | 2.0 | 1.2
  Erythema_Mild (n=191, 95, 99, 582) | 18.3 | 22.1 | 18.2 | 16.0
  Erythema_Moderate (n=191, 95, 99, 582) | 2.1 | 9.5 | 11.1 | 6.4
  Erythema_Severe (n=191, 95, 99, 582) | 0 | 0 | 0 | 0.2
  Swelling_Mild (n=191, 95, 99, 582) | 1.6 | 5.3 | 9.1 | 5.0
  Swelling_Moderate (n=191, 95, 99, 582) | 0 | 3.2 | 5.1 | 1.4
  Swelling_Severe (n=191, 95, 99, 582) | 0 | 0 | 0 | 0.2

8. Secondary Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs) by Severity
Description: The percentage of participants with solicited systemic AEs of varying severity are reported. Solicited systemic AEs are defined as asthenia, fever, headache, malaise, and myalgia that occurred at least once within 14 days after either vaccination, as recorded by the participants in a diary. Participants with multiple episodes are categorized using the highest severity level. Percentages are based on the number of participants with diary data available.
Time Frame: Days 1 through 14 after each vaccination
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Group A: TDV Liquid + Placebo | Group B: TDV Liquid | Group C: TDV Liquid | Group D: TDV Lyophilized
Number analyzed (Participants) | 191 | 95 | 99 | 584
percentage of participants
  Headache_Mild | 27.2 | 26.3 | 21.2 | 23.1
  Headache_Moderate | 8.4 | 9.5 | 13.1 | 13.5
  Headache_Severe | 5.2 | 7.4 | 4.0 | 4.5
  Asthenia_Mild | 18.8 | 11.6 | 13.1 | 16.4
  Asthenia_Moderate | 5.8 | 10.5 | 10.1 | 7.9
  Asthenia_Severe | 3.1 | 1.1 | 2.0 | 2.6
  Malaise_Mild | 17.8 | 15.8 | 15.2 | 14.0
  Malaise_Moderate | 7.3 | 9.5 | 7.1 | 8.7
  Malaise_Severe | 4.2 | 2.1 | 3.0 | 2.6
  Myalgia_Mild | 20.9 | 23.2 | 22.2 | 23.5
  Myalgia_Moderate | 7.3 | 11.6 | 6.1 | 8.4
  Myalgia_Severe | 2.1 | 4.2 | 2.0 | 1.4
  Fever_38.0 - 38.4 °C | 1.0 | 2.1 | 1.0 | 1.0
  Fever_38.5 - 38.9 °C | 0.5 | 1.1 | 0 | 0.7
  Fever_39.0 - 40.0 °C | 0 | 0 | 0 | 0
  Fever_>40 °C | 0 | 0 | 0 | 0

9. Secondary Outcome: Percentage of Participants With Any Unsolicited Adverse Events (AEs)
Description: Unsolicited AEs are any AEs that are not solicited local or systemic AEs, as defined by this study, that occurred at least once within 28 days after either vaccination. An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. The investigator assessed whether the AE was related to the study vaccination.
Time Frame: Up to Day 28 after each vaccination
Population: SS included all randomized participants who received at least 1 dose of study vaccine (or placebo), including a partial dose.
Measure: Number; unit: percentage of participants
Arm/Group | Group A: TDV Liquid + Placebo | Group B: TDV Liquid | Group C: TDV Liquid | Group D: TDV Lyophilized
Number analyzed (Participants) | 197 | 97 | 100 | 602
percentage of participants | 40.1 | 47.4 | 45.0 | 43.7

10. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) is defined as any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria.
Time Frame: Up to 6 Months after the last dose (9 months)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Group A: TDV Liquid + Placebo | Group B: TDV Liquid | Group C: TDV Liquid | Group D: TDV Lyophilized
Number analyzed (Participants) | 197 | 97 | 100 | 602
percentage of participants | 1.0 | 1.0 | 0 | 1.3

11. Secondary Outcome: Percentage of Participants With Markedly Abnormal Laboratory Values in the Safety Sub-Set
Description: Percentage of participants with markedly abnormal standard safety laboratory values collected at any time after the first vaccination.
Time Frame: Days 8, 15, 91, 97 and 104
Population: The Safety Laboratory Sub-Set included randomly chosen participants from each treatment group for whom samples for clinical safety lab tests were collected and who received at least one vaccination dose. "n" in each of the categories is the number of participants with data available at the given time-point.
Measure: Number; unit: percentage of participants
Arm/Group | Group A: TDV Liquid + Placebo | Group B: TDV Liquid | Group C: TDV Liquid | Group D: TDV Lyophilized
Number analyzed (Participants) | 121 | 61 | 64 | 405
percentage of participants
  Hemoglobin | 0 | 0 | 0 | 0.2
  Neutrophils (Abs.) | 2.5 | 0 | 0 | 0.5
  Lymphocytes (Abs.) | 0.8 | 0 | 0 | 0.5
  Eosinophils (Abs.) | 0.8 | 1.6 | 0 | 0
  Neutrophils (%) | 0.8 | 0 | 0 | 0.2
  Lymphocytes (%) | 0 | 0 | 0 | 0.5
  Eosinophils (%) | 2.5 | 1.6 | 0 | 0.5
  Platelet Count | 0 | 0 | 0 | 0.2
  Prothrombin Time | 0 | 0 | 0 | 0.7
  aPTT | 0 | 0 | 0 | 0.5
  ALT(SGPT) (n=121,61,64,404) | 3.3 | 0 | 3.1 | 1.7
  AST(SGOT) (n=121,61,64,404) | 2.5 | 0 | 1.6 | 1.5
  Alkaline Phosphatase (n=121,61,64,404) | 0.8 | 0 | 0 | 0.2
  BUN (n=121,61,64,404) | 0 | 0 | 0 | 0.2

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: 9 months. Non-Serious Adverse Events: 28 Days after each vaccination.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study vaccine.
Arm/Group | Group A: TDV Liquid + Placebo | Group B: TDV Liquid | Group C: TDV Liquid | Group D: TDV Lyophilized
Serious Adverse Events (participants affected / at risk) | 2/197 | 1/97 | 0/100 | 8/602
Other Adverse Events (participants affected / at risk) | 50/197 | 34/97 | 29/100 | 178/602
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: TDV Liquid + Placebo (N=197) | Group B: TDV Liquid (N=97) | Group C: TDV Liquid (N=100) | Group D: TDV Lyophilized (N=602)
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral artery occlusion (Nervous system disorders) | 0 | 0 | 0 | 1
Cervical cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Complex partial seizures (Nervous system disorders) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hepatitis C (Infections and infestations) | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Temporal lobe epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: TDV Liquid + Placebo (N=197) | Group B: TDV Liquid (N=97) | Group C: TDV Liquid (N=100) | Group D: TDV Lyophilized (N=602)
Injection site erythema (General disorders) | 10 | 6 | 10 | 41
Injection site pain (General disorders) | 5 | 6 | 2 | 25
Headache (Nervous system disorders) | 8 | 3 | 0 | 22
Injection site pruritus (General disorders) | 5 | 4 | 7 | 19
Nausea (Gastrointestinal disorders) | 4 | 2 | 0 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 5
Fatigue (General disorders) | 1 | 2 | 0 | 8
Injection site discolouration (General disorders) | 1 | 1 | 3 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 6
Gastroenteritis (Infections and infestations) | 1 | 4 | 0 | 5
Laceration (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 10 | 3 | 2 | 23
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 6
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 10
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 2 | 0 | 5
Vomiting (Gastrointestinal disorders) | 4 | 2 | 0 | 11
Injection site swelling (General disorders) | 0 | 2 | 1 | 8
Nasopharyngitis (Infections and infestations) | 3 | 0 | 3 | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.